CLINICAL TRIAL: NCT05825417
Title: A Multicentre Randomised Cross-over Trial of Disease Specific Therapy in Patients With Pulmonary Arterial Hypertension (PAH) Implanted With Pulmonary Artery Pressure and Cardiac Rhythm Monitoring Devices (CardioMEMS/ConfirmRx)
Brief Title: Pulmonary Hypertension: Intensification and Personalisation of Combination Rx
Acronym: PHoenix
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Glasgow (Other); University of Sheffield (Other); University of Newcastle Upon-Tyne (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STH21653; MR/W026279/1 (Other Grant/Funding Number: UKRI Medical Research Council); 325120 (Other: IRAS)
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: remote monitoring; therapeutic development; personalised medicine
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag; riociguat

STUDY DESIGN:
Intervention Model Description: 2x2 crossover study in which the effects of adding an oral drug targeting the prostacyclin pathway and the switching of PDE5i to sGCS will be examined following 12-weeks on treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm A (selexipag/riociguat) (Active Comparator): Baseline - established PDE/ERA therapy Week 1 - initiate OPA (PDE/ERA/OPA therapy) Weeks 2-12 - uptitration of OPA to maximal therapy (PDE/ERA/OPA therapy) Weeks 13-14 - reduce OPA (PDE/ERA/OPA therapy) Week 15 - washout OPA (PDE/OPA therapy) Week 16 - washout PDE (ERA therapy) Week 17 - initiate sGCS (ERA/sGCS therapy) Weeks 18-27 - uptitration of sGCS to maximal therapy (ERA/sGCS therapy)
  Interventions: Drug: Selexipag; Drug: Riociguat; Device: CardioMEMS pulmonary artery pressure monitor; Device: Confirm Rx
- Arm B (riociguat/selexipag) (Active Comparator): Baseline - established PDE/ERA therapy Week 1 - washout PDE (ERA therapy only) Week 2 - initiate sGCS (ERA/sGCS therapy) Weeks 3-12 - uptitration of sGCS to maximal therapy (ERA/sGCS therapy) Week 13 - reduce sGCS (ERA/sGCS therapy) Week 14 - reduce and washout sGCS (ERA therapy) Week 15 - initiate PDE (PDE/ERA therapy) Week 16 - initiate OPA (PDE/ERA/OPA therapy) Weeks 17-27 - uptitration of OPA to maximal therapy (PDE/ERA/OPA therapy)
  Interventions: Drug: Selexipag; Drug: Riociguat; Device: CardioMEMS pulmonary artery pressure monitor; Device: Confirm Rx

INTERVENTIONS:
Drug: Selexipag — If Arm A - Up-titration to maximum tolerated dose followed by de-escalation If Arm B - Up-titration to maximum tolerated dose followed by observation, modification or transition at discretion of responsible care team where necessary.
  Other Names: Uptravi; oral prostacyclin IP receptor agonist (OPA)
Drug: Riociguat — If Arm A - Up-titration to maximum tolerated dose followed by de-escalation If Arm B - Up-titration to maximum tolerated dose followed by observation, modification or transition at discretion of responsible care team where necessary.
  Other Names: Adempas; soluble guanylate cyclase stimulator (sGCS)
Device: CardioMEMS pulmonary artery pressure monitor — Implantation and remote monitoring established with patient initiated daily readings
Device: Confirm Rx — Implantation and remote monitoring established with automated daily readings / downloads

SUMMARY:
The goal of this clinical trial is to evaluate the capacity of implantable/remote technology for early evaluation of drug therapies in patients with pulmonary arterial hypertension (PAH). The main question it aims to answer is whether structured changes in clinical therapy will be detectable using implanted regulatory approved devices. Participants will will be implanted with approved medical devices and will enter into a study of approved drugs to assess physiology, activity and patient reported quality-of-life (QoL) outcomes. Researchers will compare two therapeutic strategies in each individual patient to see if the study design provides enough evidence to personalise drug treatment plans

DETAILED DESCRIPTION:
In this study, patients established on guideline recommended therapy will be implanted with devices and remote monitoring established. Patients will then enter into a 2x2 crossover study of approved drugs during which standard clinical investigations will be undertaken at baseline and maximal therapy on each drug. The cross-over design will provide multiple increases and decreases of drugs known to alter haemodynamics and 6MWT. The study is powered to detect improvement in right ventricular stroke volume measured by MRI from baseline to maximal therapy for each drug. It will then be established if changes in remote monitored measures provide an early indication of clinical efficacy when compared to the MRI, haemodynamics, NTproBNP and 6MWT made at 12-weeks. Remote measurement of haemodynamics during the two periods of de-escalation will inform understanding of physiology and inform clinical practice. The comparison of the two therapeutic strategies in individual patients in one study will facilitate novel clinical study designs and provide evidence for data-driven personalised medicine in the area.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Age 18-80 years
* PAH which is idiopathic, heritable or associated with drugs, toxins or connective tissue disease
* Stable PAH therapeutic regime comprising any combination of ERA and PDE5i for at least 1 month prior to screening (unless unable to tolerate therapy)
* WHO functional class III
* Resting mPAP ≥20 mmHg, pulmonary capillary wedge pressure ≤15 mmHg, pulmonary vascular resistance ≥2 Wood Units measured by right heart catheterisation at time of diagnosis
* 6MWT >50m at entry
* Estimated glomerular filtration rate (eGFR)>30 ml/min/1.73 m² at entry (Appendix C)
* Inadequate treatment response (clinically determined)

Exclusion Criteria:

* Unable to provide informed consent
* Pregnancy
* Unprovoked pulmonary embolism (at any time)
* Acute infection at time of screening (rescreening is permitted)
* PAH due to human immunodeficiency virus, portal hypertension, schistosomiasis, congenital heart disease
* Pulmonary hypertension due to left heart, lung, thromboembolic or unclear/multifactorial disease (Group II-V)
* Unable to tolerate aspirin or P2Y12 inhibitor
* Hypersensitivity to selexipag or riociguat
* Clinically-significant renal disease (eGFR≤30 ml/min/1.73m2)
* Anaemia (haemoglobin <10 g/dl)
* Left-sided heart disease and/or clinically significant cardiac disease, including but not limited to any of the following: aortic or mitral valve disease greater than mild aortic insufficiency; mild aortic stenosis; mild mitral stenosis; or moderate mitral regurgitation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Right Ventricular Stroke Volume (RVSV) flow on each therapy measured by MRI RSVS (flow) on each therapy measured by MRI | Baseline to Week 12
  This provides a robust, objective assessment of clinical efficacy which, if met, will mean that a change in therapy has provided a clinically meaningful change in physiology

SECONDARY OUTCOMES:
Haemodynamics - Total Pulmonary Resistance (TPR) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change in TPR (Woods Units) on each therapy to determine clinical efficacy
Haemodynamics - mean Pulmonary Artery Pressure (mPAP) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change in mPAP (mmHg) on each therapy to determine clinical efficacy
Haemodynamics - Cardiac Output (CO) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change in CO (L/min) on each therapy to determine clinical efficacy
Haemodynamics - Cardiac Index | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change in cardiac index (L/min/m^2) on each therapy to determine clinical efficacy
Haemodynamics - Stroke Volume (SV) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change in SV (mL) on each therapy to determine clinical efficacy
Haemodynamics - Heart Rate (HR) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change in HR (bpm) on each therapy to determine clinical efficacy
6 Minute Walk Test | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change on each therapy to determine clinical efficacy
NTpro-BNP | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change on each therapy to determine clinical efficacy
MRI - Right Ventricular Ejection Fraction (RVEF) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  RVEF (%) on each therapy to determine clinical efficacy
MRI - Right Ventricular End Systolic Volume (RVESV) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  RVESV (mL/m^2) on each therapy to determine clinical efficacy
MRI - Right Ventricular End Diastolic Volume (RVEDV) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  RVEDV (mL/m^2) on each therapy to determine clinical efficacy
MRI - Right Ventricular Stroke Volume (RVSV) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  RVSV (mL) on each therapy to determine clinical efficacy
MRI - Left Ventricular Volume Fraction (LVEF) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  LVEF (%) on each therapy to determine clinical efficacy
MRI - Left Ventricular End Systolic Volume (LVESV) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  LVESV (mL/m^2) on each therapy to determine clinical efficacy
MRI - Left Ventricular End Diastolic Volume LVEDV | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  LVEDV (mL/m^2) on each therapy to determine clinical efficacy
MRI - Left Ventricular Stroke Volume (LVSV) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  LVSV (mL) on each therapy to determine clinical efficacy
MRI - Left Ventricular Stroke Volume (LVSV) flow | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  LVSV flow on each therapy to determine clinical efficacy
Patient Reported Outcomes (PRO) - Quality of Life (QoL) (EmPHasis-10) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change of QoL score on each therapy to determine clinical efficacy. This will be done using EmPHasis-10 questionnaire (10 questions using a 0 (poor) - 5 (good) scale)
Patient Reported Outcomes (PRO) - Medication Compliance (PHoenix PRO) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change of medication compliance score on each therapy to determine clinical efficacy. This will be done using PHoenix PRO questionnaire (10 questions using a 0 (poor) - 5 (good) scale)
Patient Reported Outcomes (PRO) - Medication Side Effects | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change of medication side effects on each therapy to determine clinical efficacy. This will be done using PHoenix Medication side effects questionnaires (4 Yes/No or Better/Worse style questions)
Patient Reported Outcomes (PRO) - Depression symptoms (GAD-2/7) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change of depression symptoms on each therapy to determine clinical efficacy. This will be done using the GAD-2/7 questionnaire (2 screening questions to determine if symptoms present. If present, 7 additional questions to determine level of depression using a 0 (not at all) - 3 (nearly every day) scale)
Patient Reported Outcomes (PRO) - Anxiety symptoms (PHQ-2/9) | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change of anxiety symptoms on each therapy to determine clinical efficacy. This will be done using the PHQ-2/9 questionnaire (2 screening questions to determine if symptoms present. If present, 9 additional questions to determine level of anxiety using a 0 (not at all) - 3 (nearly every day) scale)
WHO functional class | From baseline and area under the curve to 4 weeks, 8 weeks and 12 weeks
  Change on each therapy to determine clinical efficacy. Functional assessment of PAH will be made according to the WHO classification system: Class I - Patients with PAH without limitation of physical activity. Ordinary physical activity does not cause increased dyspnoea or fatigue, chest pain, or near syncope / Class II - Patients with PAH resulting in slight limitation of physical activity. No discomfort at rest. Normal physical activity causes increased dyspnoea or fatigue, chest pain, or near syncope / Class III - Patients with PAH resulting in marked limitation of physical activity. There is no discomfort at rest. Less than ordinary activity causes increased dyspnoea or fatigue, chest pain, or near syncope / Class IV - Patients with PAH with inability to carry out any physical activity without discomfort. Indications of manifest right heart failure. Dyspnoea and/or fatigue may even be present at rest. Discomfort is increased by the least physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rothman, MD / PhD, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Research samples will be transferred to the Sheffield Biorepository with no identifiable personal data.
  Data will be collected and hosted and processed by University of Oxford (data supplier). Authorised data originators include, but are not limited to PIs and delegated staff; Participants; and Core Imaging Laboratory. The trial manager will lead the data verification process. Remote monitoring data will be managed through the Merlin.net system (Device supplier - Abbott). Pseudonymised data will then be transferred, held, analysed and archived securely at the University of Glasgow (processor). Data will also be transferred to the University of Sheffield and Newcastle University (processor) for study analysis.
  The University of Sheffield shall own all right, title and interest in and to all of the University of Sheffield Data. For the purposes of the Data Protection Legislation, Sheffield Teaching Hospitals (sponsor) is the Data Controller.

REFERENCES:
- [Background] Swift AJ, Wilson F, Cogliano M, Kendall L, Alandejani F, Alabed S, Hughes P, Shahin Y, Saunders L, Oram C, Capener D, Rothman A, Garg P, Johns C, Austin M, Macdonald A, Pickworth J, Hickey P, Condliffe R, Cahn A, Lawrie A, Wild JM, Kiely DG. Repeatability and sensitivity to change of non-invasive end points in PAH: the RESPIRE study. Thorax. 2021 Oct;76(10):1032-1035. doi: 10.1136/thoraxjnl-2020-216078. Epub 2021 Feb 25. PMID 33632769